CLINICAL TRIAL: NCT00128258
Title: Phase 1 Study: Autologous/Allogeneic Bone Marrow Progenitor Cell Treatment for Heart Failure
Brief Title: Autologous/Allogeneic Progenitor Stem Cell Therapy for Congestive Heart Failure
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study no longer at pittsburgh
Sponsor: Amit, Patel N, M.D. (Other)
Responsible Party: Principal Investigator, Amit N. Patel MD MS, Director, Amit, Patel N, M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #:0504126
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure, Congestive
Keywords: Stem Cell; Heart Failure; Bone Marrow
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- open (Experimental): open treatment
  Interventions: Procedure: Injection of bone marrow cells in the heart; Biological: Biological bone marrow cell therapy

INTERVENTIONS:
Procedure: Injection of bone marrow cells in the heart — Biological implant into the heart
Biological: Biological bone marrow cell therapy — Biological implant into the heart

SUMMARY:
This research study is being performed to find out more information about the safety and effectiveness of injecting bone marrow progenitor cells (BMPCs) from one's own hip bone into one's heart muscle. The BMPCs are the cells from which the different types of blood and other cells grow.

In patients with heart failure, the heart muscle does not pump well. Over a period of years, this continues to get worse until the patient dies of heart failure. The investigators are trying to find out if the injection of these BMPCs can make a change in the functioning of these areas of the heart muscle. Data from studies around the world have suggested that when patients with heart failure receive these cells by direct injection into their hearts they show signs of recovered heart function, however, there has been no evidence from actual studies of the cells of the patient's hearts to show how this process works. It is the investigator's plan to inject an eligible participant's heart with cells that are from one's own bone marrow during an operation to receive a ventricular assist device (VAD) or partial artificial heart and then to study the function of the heart while awaiting a heart transplant. The investigators will then examine the heart after it has been removed as part of the regular heart transplant operation for any microscopic changes (changes too small to be seen by the unaided eye but large enough to be studied under a microscope) at the site where the cells are injected. Participants will have no change in the chances of receiving a heart transplant by agreeing to participate in this study. There will also be no delay in receiving a VAD operation while waiting to participate in this study. This Phase I study has been cleared by the Food and Drug Administration (FDA) to enroll and treat patients. The Center for Biologics Evaluation and Research Investigational New Drug number (IND BB #) is 12304. (A Phase I trial is a research study using techniques or products in the first-stage or for the first time in human subjects).

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years.
* Congestive heart failure with ejection fraction <= 35.
* Candidates for ventricular device placement as a bridge to transplant.
* Serum bilirubin, SGOT and SGPT <= 2.5 times the upper level of normal.
* Serum creatinine < 2.0 times normal or no dialysis.
* New York Heart Association (NYHA) performance status > 3.
* Negative pregnancy test (in women with childbearing potential).

Exclusion Criteria:

* Pregnant or breastfeeding women.
* History of prior radiation exposure.
* History of bone marrow disorder.
* History of abnormal bleeding or clotting.
* History of liver cirrhosis.
* Inability to obtain 1 x 10^6 CD 34+ cells after bone marrow processing.
* Acute myocardial infarction < 6 days from acute event.
* Prior malignancy in the 5 years before treatment in this study (other than curatively treated carcinoma in-situ of the cervix or non-melanoma skin cancer).
* Inability or unwillingness to comply with the treatment protocol, follow-up, research tests, or give consent.
* Eligible for destination ventricular assist device placement.
* Unable to have 250cc bone marrow harvested.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-05-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Heart function at 3 months after implant | 3 months

SECONDARY OUTCOMES:
Toxicity | 3 months